CLINICAL TRIAL: NCT03912493
Title: The Effectiveness of Game-Based Virtual Reality Approach in Patients With Subacromial Impingement Syndrome
Brief Title: Virtual Reality Approach in Subacromial Impingement Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29.11.2016/36
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Shoulder Impingement Syndrome; Virtual Reality; Rehabilitation; Subacromial Impingement Syndrome
Keywords: Subacromial Impingement Syndrome; Physiotherapy and Rehabilitation; Virtual Reality; Technologic Rehabilitation
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Number of participants in this group is anticipated to be 20. Conventional physiotherapy and rehabilitation methods will be applied to this group. The conventional program includes the application of Transcutaneous Electrical Nerve Stimulation (TENS), cold pack, therapeutic ultrasound, Codman Exercises, Wand exercises, shoulder wheel exercises, finger ladder exercises, strengthening exercises with elastic band and capsule stretching.
  Interventions: Other: Conventional Physiotherapy and Rehabilitation
- Study Group (Active Comparator): Number of participants in this group is anticipated to be 20. Participants in this group will be receiving conventional physiotherapy and rehabilitation methods and 10 minutes of exercise with the game-based virtual reality system (USE-IT). In the USE-IT system two games will be played for 5 minutes each.
  Interventions: Device: Game Based Virtual Reality Exercises; Other: Conventional Physiotherapy and Rehabilitation

INTERVENTIONS:
Device: Game Based Virtual Reality Exercises — A game-based virtual reality device named USE-IT will be added to the rehabilitation program. USE-IT is a technological rehabilitation system designed by the Department of Physiotherapy and Rehabilitation at Hacettepe University. It is a smart gaming device which has been used in patients who suffer from movement loss in their upper extremities due to various neurological and orthopedic reasons.
  Arms: Study Group
Other: Conventional Physiotherapy and Rehabilitation — The conventional physiotherapy and rehabilitation program includes the application of Transcutaneous Electrical Nerve Stimulation (TENS), cold pack, therapeutic ultrasound, Codman Exercises, Wand exercises, shoulder wheel exercises, finger ladder exercises, strengthening exercises with elastic band and capsule stretching.

SUMMARY:
The aim of our study is to investigate the effects of game-based virtual reality exercise added to conventional physiotherapy and rehabilitation program in patients with Subacromial Impingement Syndrome (SIS). In order to evaluate its effectiveness, assessment of pain, range of motion and disability will be applied.

DETAILED DESCRIPTION:
Subacromial Impingement Syndrome (SIS) is the result of contraction of the structures passing through the subacromial area. Problems in upper limb function in people with SIS adversely affect quality of life and functional independence of the patients. Recovery of restricted daily life functions (such as dressing, personal care, eating and body care) is one of the main goals of physiotherapy and rehabilitation in SIS and currently, conventional physiotherapy and rehabilitation methods are most commonly used. The main purpose of this method is to reduce pain, increase range of motion and muscle strength. With the developing technology various virtual reality applications have begun to take place in physiotherapy and rehabilitation programs recently. These virtual reality applications are used to motivate the patient and keep their interest in the rehabilitation. In addition, the diversity of virtual reality applications is increasing day by day so that participation of the patients and the interest in the treatment can be increased. Various measurements of the user's performance can be transferred to the clinician simultaneously with these systems. Also for most of these systems exercise modes, difficulty and duration are programmable so that the training sessions can be varied. The aim of our study is to investigate the effects of game-based virtual reality exercises added to conventional physiotherapy and rehabilitation program in patients with SIS.

ELIGIBILITY:
Inclusion Criteria:

* Volunteered to participate in the study
* Aged 18-65 years,

Exclusion Criteria:

* Any visual or hearing problem,
* Other neurological, orthopedic or rheumatic problems that may restrict shoulder motion or cause pain,
* Having a physical disability or uncontrolled chronic systemic disease,
* Major trauma,
* Treatment for shoulder problems within the last 6 months,
* History of epileptic attacks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in range of motion from baseline to week 4 | 4 weeks
  The range of motion of the joints in the upper extremities will be measured using the universal goniometer before and after the treatment.
Change in level of pain from baseline to week 4 | 4 weeks
  Level of Pain will be assessed with Visual Analogue Scale (VAS). It is widely used among the methods of measuring the severity of pain. Scale is a 10 cm ruler, participants will mark the level of pain between 0-10 cm, 0 would means ''no pain'' and 10 would means ''worst possible pain''.
Change in disability of the upper extremity from baseline to week 4 | 4 weeks
  Disability of the upper extremities will be assessed with 'The Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire'. It is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The questionnaire was designed to help describe the disability experienced by people with upper-limb disorders and also to monitor changes in symptoms and function over time.
Change in quality of shoulder function from baseline to week 4 | 4 weeks
  Quality of function of the shoulder will be assessed with Constant-Murley Score. It is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. Pain (15 points), daily living activities (20 points), active range of motion (40 points) and force (25 points) parameters, including a total of 100 points system. The total Constant score is classified as excellent (30 <), good (21 - 30), medium (11 - 20) and weak (<11).
Change in muscle strength from baseline to week 4 | 4 weeks
  The muscle strength of shoulder flexion, abduction, adduction, external and internal rotation movements will be evaluated by using the Baseline Push-Pull (New York) dynamometer. Results will be calculated in kg (1 lb = 0.454 kg). The patient's arm will be stabilized and the patient will be asked to show maximum resistance within 2 sec against the dynamometer placed and then hold it for 5 seconds at this position and power. The measurement will be repeated twice and recorded with the average of these two values.
Change in pain threshold from baseline to week 4 | 4 weeks
  The pain threshold will be measured with a digital algometer device. Algometers are devices that can be used to identify the pressure and/or force eliciting a pressure-pain threshold. It has been noted in pressure-pain threshold studies that the rate at which manual force is applied should be consistent to provide the greatest reliability.
Change in proprioception from baseline to week 4 | 4 weeks
  Proprioception will be evaluated with 'Marmara Visual Auditory Joint Education Device (MarVAJED) which was developed by the Faculty of Health Sciences of Marmara University, Istanbul. This device evaluates motion deficits of joints, analyzes joint position sense, provides biofeedback support to increase joint control and also directs to controlled exercises. It analyzes the motion of the joint with the help of small sensors and transfers the data obtained to the mobile phone, tablet or computer.
Change in kinesiophobia from baseline to week 4 | 4 weeks
  In the assessment of kinesiophobia 'Tampa Kinesiophobia Scale (TKS)' will be used. It is a 17 item questionnaire used to assess the subjective rating of kinesiophobia or fear of movement. The scale is based on the model of fear avoidance, fear of work related activities, fear of movement and fear of re-injury.
Satisfaction of the Treatment | 4 weeks
  An objective test that evaluates the satisfaction of the patient from pain status, functionality, treatment and physiotherapist after treatment will be assessed with 4 questions, and each question is given a score of 0-10 using the VAS scale. 0 means ''I am not satisfied at all'', 10 means ''I am very satisfied''.

CONTACTS AND LOCATIONS:
Overall Officials: Berivan Beril KILIC, MSc, PT, Principal Investigator — Marmara University Institute of Health Sciences; Zübeyir SARI, Assoc Prof, Study Director — Marmara University Faculty of Health Sciences
Locations (1):
- Cadde Tıp Merkezi - Cadde Medical Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrews AW, Thomas MW, Bohannon RW. Normative values for isometric muscle force measurements obtained with hand-held dynamometers. Phys Ther. 1996 Mar;76(3):248-59. doi: 10.1093/ptj/76.3.248. PMID 8602410
- [Background] Arman N, Tarakci E, Tarakci D, Kasapcopur O. Effects of Video Games-Based Task-Oriented Activity Training (Xbox 360 Kinect) on Activity Performance and Participation in Patients With Juvenile Idiopathic Arthritis: A Randomized Clinical Trial. Am J Phys Med Rehabil. 2019 Mar;98(3):174-181. doi: 10.1097/PHM.0000000000001001. PMID 30020092
- [Background] Bao X, Mao Y, Lin Q, Qiu Y, Chen S, Li L, Cates RS, Zhou S, Huang D. Mechanism of Kinect-based virtual reality training for motor functional recovery of upper limbs after subacute stroke. Neural Regen Res. 2013 Nov 5;8(31):2904-13. doi: 10.3969/j.issn.1673-5374.2013.31.003. PMID 25206611
- [Background] Burdea GC. Virtual rehabilitation--benefits and challenges. Methods Inf Med. 2003;42(5):519-23. PMID 14654886
- [Background] Chen CC. Multimedia virtualized environment for shoulder pain rehabilitation. J Phys Ther Sci. 2016 Apr;28(4):1349-54. doi: 10.1589/jpts.28.1349. Epub 2016 Apr 28. PMID 27190481
- [Background] Chiu HC, Ada L, Lee HM. Upper limb training using Wii Sports Resort for children with hemiplegic cerebral palsy: a randomized, single-blind trial. Clin Rehabil. 2014 Oct;28(10):1015-24. doi: 10.1177/0269215514533709. Epub 2014 May 21. PMID 24849793
- [Background] de Witte PB, Nagels J, van Arkel ER, Visser CP, Nelissen RG, de Groot JH. Study protocol subacromial impingement syndrome: the identification of pathophysiologic mechanisms (SISTIM). BMC Musculoskelet Disord. 2011 Dec 14;12:282. doi: 10.1186/1471-2474-12-282. PMID 22168667
- [Background] Foley L, Maddison R. Use of active video games to increase physical activity in children: a (virtual) reality? Pediatr Exerc Sci. 2010 Feb;22(1):7-20. doi: 10.1123/pes.22.1.7. PMID 20332536
- [Background] Hanratty CE, McVeigh JG, Kerr DP, Basford JR, Finch MB, Pendleton A, Sim J. The effectiveness of physiotherapy exercises in subacromial impingement syndrome: a systematic review and meta-analysis. Semin Arthritis Rheum. 2012 Dec;42(3):297-316. doi: 10.1016/j.semarthrit.2012.03.015. Epub 2012 May 18. PMID 22607807
- [Background] Iosa M, Morone G, Fusco A, Castagnoli M, Fusco FR, Pratesi L, Paolucci S. Leap motion controlled videogame-based therapy for rehabilitation of elderly patients with subacute stroke: a feasibility pilot study. Top Stroke Rehabil. 2015 Aug;22(4):306-16. doi: 10.1179/1074935714Z.0000000036. Epub 2015 Feb 25. PMID 26258456
- [Background] Lanningham-Foster L, Foster RC, McCrady SK, Jensen TB, Mitre N, Levine JA. Activity-promoting video games and increased energy expenditure. J Pediatr. 2009 Jun;154(6):819-23. doi: 10.1016/j.jpeds.2009.01.009. Epub 2009 Mar 25. PMID 19324368
- [Background] MacIntosh A, Lam E, Vigneron V, Vignais N, Biddiss E. Biofeedback interventions for individuals with cerebral palsy: a systematic review. Disabil Rehabil. 2019 Oct;41(20):2369-2391. doi: 10.1080/09638288.2018.1468933. Epub 2018 May 12. PMID 29756481
- [Background] Matijevic V, Secic A, Masic V, Sunic M, Kolak Z, Znika M. Virtual reality in rehabilitation and therapy. Acta Clin Croat. 2013 Dec;52(4):453-7. PMID 24696995
- [Background] Meeusen R, Lievens P. The use of cryotherapy in sports injuries. Sports Med. 1986 Nov-Dec;3(6):398-414. doi: 10.2165/00007256-198603060-00002. PMID 3538270
- [Background] Michener LA, Walsworth MK, Burnet EN. Effectiveness of rehabilitation for patients with subacromial impingement syndrome: a systematic review. J Hand Ther. 2004 Apr-Jun;17(2):152-64. doi: 10.1197/j.jht.2004.02.004. PMID 15162102
- [Background] Millar AL, Lasheway PA, Eaton W, Christensen F. A retrospective, descriptive study of shoulder outcomes in outpatient physical therapy. J Orthop Sports Phys Ther. 2006 Jun;36(6):403-14. doi: 10.2519/jospt.2006.2101. PMID 16776489
- [Background] Monge Pereira E, Molina Rueda F, Alguacil Diego IM, Cano de la Cuerda R, de Mauro A, Miangolarra Page JC; CONSOLIDER-Ingenio 2010. Use of virtual reality systems as proprioception method in cerebral palsy: clinical practice guideline. Neurologia. 2014 Nov-Dec;29(9):550-9. doi: 10.1016/j.nrl.2011.12.004. Epub 2012 Feb 17. English, Spanish. PMID 22341675
- [Background] Othman A, Taylor G. Is the constant score reliable in assessing patients with frozen shoulder? 60 shoulders scored 3 years after manipulation under anaesthesia. Acta Orthop Scand. 2004 Feb;75(1):114-6. doi: 10.1080/00016470410001708230. PMID 15022820
- [Background] Palacios-Cena D, Ortiz-Gutierrez RM, Buesa-Estellez A, Galan-Del-Rio F, Cachon Perez JM, Martinez-Piedrola R, Velarde-Garcia JF, Cano-DE-LA-Cuerda R. Multiple sclerosis patients' experiences in relation to the impact of the kinect virtual home-exercise programme: a qualitative study. Eur J Phys Rehabil Med. 2016 Jun;52(3):347-55. Epub 2016 Feb 17. PMID 26883340
- [Background] Parsons TD, Rizzo AA, Rogers S, York P. Virtual reality in paediatric rehabilitation: a review. Dev Neurorehabil. 2009 Aug;12(4):224-38. doi: 10.1080/17518420902991719. PMID 19842822
- [Background] Pekyavas NO, Ergun N. Comparison of virtual reality exergaming and home exercise programs in patients with subacromial impingement syndrome and scapular dyskinesis: Short term effect. Acta Orthop Traumatol Turc. 2017 May;51(3):238-242. doi: 10.1016/j.aott.2017.03.008. Epub 2017 Apr 24. PMID 28446376
- [Background] Philips HC. Avoidance behaviour and its role in sustaining chronic pain. Behav Res Ther. 1987;25(4):273-9. doi: 10.1016/0005-7967(87)90005-2. No abstract available. PMID 3662989
- [Background] Rubin BD, Kibler WB. Fundamental principles of shoulder rehabilitation: conservative to postoperative management. Arthroscopy. 2002 Nov-Dec;18(9 Suppl 2):29-39. doi: 10.1053/jars.2002.36507. No abstract available. PMID 12426529
- [Background] Skjaeret N, Nawaz A, Morat T, Schoene D, Helbostad JL, Vereijken B. Exercise and rehabilitation delivered through exergames in older adults: An integrative review of technologies, safety and efficacy. Int J Med Inform. 2016 Jan;85(1):1-16. doi: 10.1016/j.ijmedinf.2015.10.008. Epub 2015 Oct 28. PMID 26559887
- [Background] Shin JH, Ryu H, Jang SH. A task-specific interactive game-based virtual reality rehabilitation system for patients with stroke: a usability test and two clinical experiments. J Neuroeng Rehabil. 2014 Mar 6;11:32. doi: 10.1186/1743-0003-11-32. PMID 24597650
- [Background] Sin H, Lee G. Additional virtual reality training using Xbox Kinect in stroke survivors with hemiplegia. Am J Phys Med Rehabil. 2013 Oct;92(10):871-80. doi: 10.1097/PHM.0b013e3182a38e40. PMID 24051993
- [Background] Sluka KA, Bjordal JM, Marchand S, Rakel BA. What makes transcutaneous electrical nerve stimulation work? Making sense of the mixed results in the clinical literature. Phys Ther. 2013 Oct;93(10):1397-402. doi: 10.2522/ptj.20120281. Epub 2013 May 2. PMID 23641031
- [Background] Smith CK, Silverstein BA, Fan ZJ, Bao S, Johnson PW. Psychosocial factors and shoulder symptom development among workers. Am J Ind Med. 2009 Jan;52(1):57-68. doi: 10.1002/ajim.20644. PMID 18942665
- [Background] Senbursa G, Baltaci G, Atay OA. The effectiveness of manual therapy in supraspinatus tendinopathy. Acta Orthop Traumatol Turc. 2011;45(3):162-7. doi: 10.3944/AOTT.2011.2385. PMID 21765229
- [Background] Tarakci D, Ozdincler AR, Tarakci E, Tutuncuoglu F, Ozmen M. Wii-based Balance Therapy to Improve Balance Function of Children with Cerebral Palsy: A Pilot Study. J Phys Ther Sci. 2013 Sep;25(9):1123-7. doi: 10.1589/jpts.25.1123. Epub 2013 Oct 20. PMID 24259928
- [Background] Gunay Ucurum S, Kaya DO, Kayali Y, Askin A, Tekindal MA. Comparison of different electrotherapy methods and exercise therapy in shoulder impingement syndrome: A prospective randomized controlled trial. Acta Orthop Traumatol Turc. 2018 Jul;52(4):249-255. doi: 10.1016/j.aott.2018.03.005. Epub 2018 Apr 25. PMID 29703659
- [Background] van der Windt DAWM, van der Heijden GJMG, van den Berg SGM, Ter Riet G, de Winter AF, Bouter LM. Ultrasound therapy for musculoskeletal disorders: a systematic review. Pain. 1999 Jun;81(3):257-271. doi: 10.1016/S0304-3959(99)00016-0. PMID 10431713
- [Background] Yeldan I, Cetin E, Ozdincler AR. The effectiveness of low-level laser therapy on shoulder function in subacromial impingement syndrome. Disabil Rehabil. 2009;31(11):935-40. doi: 10.1080/09638280802377985. PMID 19031167
- [Background] Weichert F, Bachmann D, Rudak B, Fisseler D. Analysis of the accuracy and robustness of the leap motion controller. Sensors (Basel). 2013 May 14;13(5):6380-93. doi: 10.3390/s130506380. PMID 23673678
- [Background] Weiss PL, Tirosh E, Fehlings D. Role of virtual reality for cerebral palsy management. J Child Neurol. 2014 Aug;29(8):1119-24. doi: 10.1177/0883073814533007. Epub 2014 May 5. PMID 24799367
- [Background] Woollacott M, Shumway-Cook A. Attention and the control of posture and gait: a review of an emerging area of research. Gait Posture. 2002 Aug;16(1):1-14. doi: 10.1016/s0966-6362(01)00156-4. PMID 12127181

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT03912493/Prot_SAP_000.pdf